CLINICAL TRIAL: NCT06290453
Title: The Regulatory Role of miRNA 27 and Follistatin Like Protein-1 Gene in the Pathophysiology of Multiple Sclerosis Patients.
Brief Title: The Regulatory Role of miRNA 27 Follistatin Like Protein-1 Gene in Multiple Scelerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Mohammed Ali, Lecturer of medical physiology, Assiut University
Other Study IDs: AOGR
Record Dates: First submitted 2024-02-20; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Multiple sclerosis patients (MS): included 40 patients with newly discovered MS (duration of the disease is 3 years or less) and diagnosed according to the revised McDonald criteria. The patients will be recruited from the neurology department of Assiut University Hospital.
  MS patients will be further subdivided into two subgroups: 20 patients with RRMS and 20 patients with Progressive MS group.
  Interventions: Diagnostic Test: micro RNA 27- FLP1 gene expression; Diagnostic Test: The Expanded Disability Status Scale (EDSS); Diagnostic Test: Electrophysiological assessment:; Diagnostic Test: MRI examination MRI brain:
- Control (C): Group II: included 20 healthy individuals who will be age- and sex-matched as a control group, with no history of any neurological or autoimmune disease.
  Interventions: Diagnostic Test: micro RNA 27- FLP1 gene expression

INTERVENTIONS:
Diagnostic Test: micro RNA 27- FLP1 gene expression — From each participant, 2 mL of blood will be drawn and store at 25-degree C. The expression of miRNA-27 and FLP1 gene will be measured using real time PCR.
  Relative expression values will be normalised to the housekeeping gene GAPDH. The comparative cycle threshold (Ct) approach will be used to measure the relative expression of miRNA 27 and FLP1 gene. Then, using the equation -ΔΔCT, the fold change of each gene will be determined
Diagnostic Test: The Expanded Disability Status Scale (EDSS) — The Expanded Disability Status Scale (EDSS) is a way of measuring how much someone is affected by their MS. Neurologists use it to monitor changes in the level of someone's disability over time. The EDSS has a range from 0 to 10.
  Zero points is normal neurological examination. 10 points shows the MS-related death cases. Patients with EDSS score up to 5 are fully ambulatory patients.
  Groups: Multiple sclerosis patients (MS)
Diagnostic Test: Electrophysiological assessment: — Electromyography and nerve conduction velocity will be performed for all MS patients.
  Groups: Multiple sclerosis patients (MS)
Diagnostic Test: MRI examination MRI brain: — will be done on all MS patients to detect the number, the site, and the enhancement of lesions
  Groups: Multiple sclerosis patients (MS)

SUMMARY:
Multiple sclerosis (MS) is a neurodegenerative disease characterized by demyelination of the central nervous system. Young women between the ages of 20 and 40 are primarily targeted by this disabling disorder. Till now there are no sufficient mechanisms to explain the pathophysiology of multiple sclerosis.

DETAILED DESCRIPTION:
Neuroinflammation has been implicated in the initiation and progression of several central nervous system (CNS) disorders, including multiple sclerosis. Microglia and astrocytes are essential in neural development, maintenance of synaptic connections, and homeostasis in a healthy brain.

Recent researchers have discovered that microRNAs (miRNAs) contribute to the pathophysiology of MS, primarily influencing glial cells and the immune cells in the periphery. In recent years, miRNAs have become more prevalent as inflammation and demyelination process regulators in MS.

miRNAs are naturally occurring, non-coding RNA molecules (21-25 nucleotides). miRNAs play a part in the post-transcriptional regulation of gene expression and silencing of RNA. miRNAs have been discovered to control some physiological processes, as apoptosis, proliferation, differentiation, and development.

Measurement of circulating miRNAs in MS patients' peripheral blood is one of the promising approaches as it can be a non-invasive tool to explain its pathogenesis. miRNAs are remarkably stable in bodily fluids and are relatively simple to collect and quantify. Moreover, a novel approach to therapy may be based on methods that regulate the activity of miRNAs.

Several miRNAs particularly miR-27 have been reportedly involved in regulating myelination in the central nervous system. However, the role of micro RNAs in generation or progression of MS remains elusive.

Follistatin-like protein-1 (FSTL1) was first identified as a transforming growth factor β1-inducible protein. In the last decade, FSTL1 has been identified as a novel inflammatory protein. FSTL1 is a glycoprotein rich in cysteine (SPARC) family. FSTL1 is elevated in various inflammatory conditions and decreased during treatment.

Moreover, a variety of studies suggest that targeting of FSTL1 may be useful in the treatment of diseases in which inflammation plays a central role. Recent studies revealed a substantial connection between FSTL1 and micro-RNA 27 levels and demonstrated that the regulatory effects of miR-27 in some inflammatory conditions may be exerted by targeting FSTL1.

This study aims to investigate the expression patterns of miR-27 and Follistatin like 1 gene in peripheral blood samples of MS patients. As, we hypothesize that miR-27 and its target gene (FSTL1) may serve important roles in the pathogenesis of MS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MS based on the revised McDonald criteria.
2. Female patients will only be included.
3. 20- 45 years old.
4. Drug naïve.

Exclusion Criteria:

* 1. Patients with other neurodegenerative and autoimmune disorders. 2. Pregnant females. 3. Co-existing chronic hypertension, diabetes, and epilepsy 4. chronic renal or hepatic diseases

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Study subjects:
  1. Inclusion criteria:
     1. Patients diagnosed with MS based on the revised McDonald criteria.
     2. Female patients will only be included.
     3. 20- 45 years old.
     4. Drug naïve.
  2. Exclusion criteria:
     1. Patients with other neurodegenerative and autoimmune disorders.
     2. Pregnant females.
     3. Co-existing chronic hypertension, diabetes, and epilepsy
     4. Chronic renal or hepatic diseases
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
• To measure the levels of miR-27 expression and its target gene (FSTL1) in progressive MS and relapsing-remitting multiple sclerosis (RRMS) patients. | 1 month
  RNA extraction Reverse Transcription polymerase chain reaction (RT-PCR) analysis:

SECONDARY OUTCOMES:
To correlate the levels of expression of miR-27 expression and its target gene (FSTL1) relative to the severity of symptoms of MD patients. | 1 month
  Statistical analysis: Pearson correlation for parametric data, spearman correlation for non-parametric data.

REFERENCES:
- [Result] Chaly Y, Marinov AD, Oxburgh L, Bushnell DS, Hirsch R. FSTL1 promotes arthritis in mice by enhancing inflammatory cytokine/chemokine expression. Arthritis Rheum. 2012 Apr;64(4):1082-8. doi: 10.1002/art.33422. Epub 2011 Oct 17. PMID 22006268
- [Result] Chen L, Lu Q, Chen J, Feng R, Yang C. Upregulating miR-27a-3p inhibits cell proliferation and inflammation of rheumatoid arthritis synovial fibroblasts through targeting toll-like receptor 5. Exp Ther Med. 2021 Nov;22(5):1227. doi: 10.3892/etm.2021.10661. Epub 2021 Aug 27. PMID 34539823
- [Result] Mattiotti A, Prakash S, Barnett P, van den Hoff MJB. Follistatin-like 1 in development and human diseases. Cell Mol Life Sci. 2018 Jul;75(13):2339-2354. doi: 10.1007/s00018-018-2805-0. Epub 2018 Mar 29. PMID 29594389
- [Result] Pachner AR. The Neuroimmunology of Multiple Sclerosis: Fictions and Facts. Front Neurol. 2022 Feb 7;12:796378. doi: 10.3389/fneur.2021.796378. eCollection 2021. PMID 35197914
- [Result] Shi DL, Shi GR, Xie J, Du XZ, Yang H. MicroRNA-27a Inhibits Cell Migration and Invasion of Fibroblast-Like Synoviocytes by Targeting Follistatin-Like Protein 1 in Rheumatoid Arthritis. Mol Cells. 2016 Aug 31;39(8):611-8. doi: 10.14348/molcells.2016.0103. Epub 2016 Aug 8. PMID 27498552
- [Result] Sun M, You H, Hu X, Luo Y, Zhang Z, Song Y, An J, Lu H. Microglia-Astrocyte Interaction in Neural Development and Neural Pathogenesis. Cells. 2023 Jul 27;12(15):1942. doi: 10.3390/cells12151942. PMID 37566021
- [Result] Zheleznyakova GY, Piket E, Needhamsen M, Hagemann-Jensen M, Ekman D, Han Y, James T, Khademi M, Al Nimer F, Scicluna P, Huang J, Kockum I, Faridani OR, Olsson T, Piehl F, Jagodic M. Small noncoding RNA profiling across cellular and biofluid compartments and their implications for multiple sclerosis immunopathology. Proc Natl Acad Sci U S A. 2021 Apr 27;118(17):e2011574118. doi: 10.1073/pnas.2011574118. PMID 33879606
- [Result] Yang J, Hamade M, Wu Q, Wang Q, Axtell R, Giri S, Mao-Draayer Y. Current and Future Biomarkers in Multiple Sclerosis. Int J Mol Sci. 2022 May 24;23(11):5877. doi: 10.3390/ijms23115877. PMID 35682558
- [Result] Tsuchikawa Y, Kamei N, Sanada Y, Nakamae T, Harada T, Imaizumi K, Akimoto T, Miyaki S, Adachi N. Deficiency of MicroRNA-23-27-24 Clusters Exhibits the Impairment of Myelination in the Central Nervous System. Neural Plast. 2023 Mar 22;2023:8938674. doi: 10.1155/2023/8938674. eCollection 2023. PMID 37006814